CLINICAL TRIAL: NCT01778647
Title: Omega-3 Fatty Acids as an Adjunctive Therapy for Stimulants in Children With ADHD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Co-Investigators left the Institution.
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Administration Director, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LVZ113607; 09/06/VA05 (Other: Maimonides Medical Center); NCT01233856 (obsolete NCT alias)
Record Dates: First submitted 2010-09-30; First posted 2013-01-29 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Omega- 3 Fatty acids; CGI; Conners rating scale; Stimulants
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Central Nervous System Stimulants; Omacor; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stimulants plus Lovaza (Experimental): Usual dose of stimulant plus Lovaza (prescription Omega-3 fatty acids) at a dose of 1800 mg daily.
  Interventions: Dietary Supplement: Stimulants plus Lovaza
- Stimulants plus placebo (Placebo Comparator): Usual dose of stimulants plus placebo(corn oil), which will be given to the patients by MMC's pharmacy.
  Interventions: Drug: Stimulants plus placebo

INTERVENTIONS:
Dietary Supplement: Stimulants plus Lovaza — Patients randomized to stimulants plus Lovaza (Omega-3 fatty acids). Treated and evaluated for up to 16 weeks. Conners and CGI scales filled out by parents, teachers and evaluators on each visit
  Other Names: Lovaza plus stimulants
  Arms: Stimulants plus Lovaza
Drug: Stimulants plus placebo — Patients randomized to usual dose of stimulants plus placebo. Patients evaluated for up to 16 weeks. Conners rating scales and CGI filled out by evaluators, parents and teachers.
  Other Names: Sugar pill plus stimulants
  Arms: Stimulants plus placebo

SUMMARY:
Multiple forms of Omega-3 Fatty acids have been used to investigate the role of this food supplement in children with Attention Deficit Hyperactivity Disorder (ADHD). No clear evidence for their role in this disorder is yet available. We will conduct a prospective, randomized, double blind, placebo controlled trial to obtain significant results regarding this question.

DETAILED DESCRIPTION:
A total of 30-150 patients or more between the ages of 6 and 15 years old with diagnosis of ADHD according to the DSM-IV and on current treatment with stimulants recruited from CAOS-MMC and the Developmental Center will be evaluated by a child psychiatrist or a resident under supervision of a child psychiatrist to make sure that the diagnosis is correct. Every child will have a Conners rating scale filled out by the parents and teachers on admission to the study. The evaluators will also fill out a Clinical Global Impression scale (CGI).

The patients will be divided in 2 groups. One group of 15 children will be randomized to continue taking the usual dose of stimulants plus placebo (corn oil), which will be given to the patients by MMC's pharmacy.

A second group of 15 patients will be randomized to receive the usual dose of stimulant plus Lovaza (prescription Omega-3 fatty acids) at a dose of 1800 mg daily.

Both groups will be initially treated for a period of 8 weeks. The patients will be re-evaluated by the investigators on week 2, 4, 6 and 8 of the study and on each evaluation the parents and teachers will fill out a Conners rating scale.

The ratings of the Conners rating scales filled for each patient will be analyzed and compared to the initial evaluation after week 8. The evaluators will also do a CGI score for every visit.

Patients that improve will be taken off the stimulants and will continue further treatment with the adjunctive therapy for a total of 4 more weeks, during this period of time they will be re-evaluated on weeks 9, 10 and 12 and Conners scales will also be filled out by the parents.

Patients who do not improve will be switched to the opposite treatment modality and will be evaluated on weeks 9, 10 and 12 also having Conners scales filled out by their parents. If any of the patients in this group improve after the switch, they will be taken off stimulants and they will be evaluated on weeks 13, 14 and 16 of the study arm.

The study will be supported by GlaxoSmithKline. This pharmaceutical company will provide the capsules and the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Children 6 to 15 years old
* Diagnosis of ADHD according to the DSM IV -TR

Exclusion Criteria:

* Children younger than 6 y/o or older than 15 y/o
* Children with other co-morbid disorders according to the DSM IV-TR
* Mentally retarded children
* Poor compliance with treatment
* Children with a diagnosis of blood clotting problems
* Children on anticoagulants
* Children with hypersensitivity to fish
* Children "In care" (CiC): Foster children or children that are not being taken care of by a biological parent or a legal guardian.
* Children who follow a kosher diet (Lovaza is not kosher)
* Pregnancy

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Conners Rating Scale for assessment of ADHD characteristics | 16 WEEKS
  Conners Rating Scales is designed to provide an overview of child and adolescent concerns and disorders, including ADHD. The survey for parents contains 80 items and 59 items for teachers. Scoring is based on a response about specific aspects of child behavior, with a low cumulative score showing less likelihood of a specific disorder. The cumulative score is called a T-score. T-scores have a mean of 50 and a standard deviation of 10. These can be converted to percentile scores. T-scores above 60 are cause for concern and have interpretive value. Interpretable scores range from a low T-score of 61 (mildly atypical) to above 70 (markedly atypical).

SECONDARY OUTCOMES:
Clinical Global Impression - Severity Scale (CGI-S) | 16 WEEKS
  The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. The CGI-Severity (CGI-S) asks the clinician one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Malloy, MD, Principal Investigator — Maimonides Medical Center; Juan D Pedraza, MD, Study Director — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Derived] Gillies D, Leach MJ, Perez Algorta G. Polyunsaturated fatty acids (PUFA) for attention deficit hyperactivity disorder (ADHD) in children and adolescents. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD007986. doi: 10.1002/14651858.CD007986.pub3. PMID 37058600